CLINICAL TRIAL: NCT07185230
Title: Atosiban in Women With Previous Implantation Failure and Abnormal Uterine Contractions Undergoing Single Blastocyst-Stage Embryo Transfer: A Randomised Triple-Blind, Placebo-Controlled Trial
Brief Title: Atosiban in Women With Previous Implantation Failure and Abnormal Uterine Contractions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Principal Investigator, He Cai, Principal investigator, Northwest Women's and Children's Hospital, Xi'an, Shaanxi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-058-02
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Infertility
Keywords: Atosiban
MeSH Terms: conditions — Infertility | interventions — atosiban

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atosiban group (Experimental): Participants allocated to the Atosiban group will be administered Atosiban
  Interventions: Drug: Atosiban
- Placebo group (Placebo Comparator): Participants allocated to the placebo group will receive saline infusions.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Atosiban — Participants allocated to the Atosiban group will be administered Atosiban (37.5 mg/5 mL, Tractocile®, Ferring Pharma, Geneva, Switzerland) as an intravenous (IV) bolus of 6·75 mg/0.9 mL in 1 minute at 30 minutes prior to the ET procedure, followed by an IV infusion at a rate of 18 mg/h for 1 hour; after 1 hour, the dose of Atosiban will be reduced to 6 mg/h, with a total dose of 37.5 mg.
  Arms: Atosiban group
Drug: Placebo Control — Participants allocated to the placebo group will receive identical-looking saline infusions for the same duration.
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the efficacy of atosiban in patients with previous pregnancy failure and abnormal uterine contractions during the peri-embryo transfer period in assisted reproductive technology. The main questions it aims to answer are:

* Does the use of atosiban in patients with a history of implantation failure and abnormal uterine contractions affect the live birth rate in single blastocyst transfer cycles (fresh or frozen-thawed embryo transfer)?
* Evaluate the differences in efficacy of atosiban regarding perinatal complications and neonatal outcomes, as well as differences in safety concerning miscarriage rates and ectopic pregnancy rates.

Researchers will compare atosiban with placebo (a similar substance containing no active medication) to determine whether atosiban is effective in improving live birth rates from single blastocyst transfer cycles (fresh or frozen-thawed embryo transfer) in patients with a history of implantation failure and abnormal uterine contractions.

* Participants allocated to the Atosiban group will be administered Atosiban (37.5 mg/5 mL, Tractocile®, Ferring Pharma, Geneva, Switzerland) as an intravenous (IV) bolus of 6·75 mg/0.9 mL in 1 minute at 30 minutes prior to the ET procedure, followed by an IV infusion at a rate of 18 mg/h for 1 hour; after 1 hour, the dose of Atosiban will be reduced to 6 mg/h, with a total dose of 37.5 mg. Participants allocated to the placebo group will receive identical-looking saline infusions for the same duration.
* One hour post-embryo transfer, all randomized participants will be invited to have a reevaluation of uterine wave patterns via ultrasound, performed by the same examiner.
* Women who had a clinical pregnancy will be subsequently contacted by nurses to document pregnancy events and outcomes at 12 and 24 weeks of gestation, completion of pregnancy, with a follow-up approximately 6 weeks post-delivery. Those participants who had a negative pregnancy test will not be followed up any further as part of this trial.

ELIGIBILITY:
Participants/eligibility criteria

Infertile women who fulfill all of the following inclusion criteria, based on the results and findings of the Atosiban 1 study are eligible for participation:

1. Scheduled for single blastocyst-stage embryo transfer, either in a fresh or frozen transfer cycle;
2. Have a history of one or more episodes of implantation failures in previous embryo transfer cycles;
3. Age between 20 and 40 years (inclusive);
4. Exhibit abnormal uterine peristalsis on transvaginal ultrasound performed on the morning of the scheduled blastocyst transfer, defined as either: high-frequency peristalsis (>4 contractions per minute), or a negative wave pattern (fundus-to-cervix direction) at any frequency.
5. Each woman could only participate in one transfer cycle.

Exclusion criteria

1. Immunologic or endocrine disorders including thyroid dysfunction, antiphospholipid syndrome, hyperprolactinemia and other severe systematic diseases (e.g., hypertension, diabetes, etc.)
2. Uterine malformations (e.g., intrauterine adhesions; unicornuate, bicornuate or septate uterus)；
3. Untreated hydrosalpinx or endometrial polyp；
4. Cycles that included in-vitro maturation or oocyte donation；
5. Prior participation in Atosiban 1 study；
6. Current participation in any other clinical trial；
7. Inability to provide informed consent to the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 792 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Live birth | After 24 weeks of gestation
  Live birth is defined as the delivery of at least one newborn who exhibits any sign of life.

SECONDARY OUTCOMES:
Biochemical pregnancy | 12 days after blastocyst transfer
  Biochemical pregnancy is defined as serum beta-human chorionic gonadotropin β-hCG> 10 IU/L 12 days after blastocyst transfer.
Clinical pregnancy | 6-8 weeks after blastocyst transfer.
  Clinical pregnancy is defined as observed gestational sac or definitive clinical signs of pregnancy observed at ultrasonography (including clinically documented ectopic pregnancy)
Ongoing pregnancy | After 12 weeks of gestation
  Ongoing pregnancy is defined as the presence of a gestational sac and fetal heartbeat after 12 weeks of gestation.
Miscarriage | before 20 weeks of gestation.
  Miscarriage is defined as spontaneous loss of an intrauterine pregnancy prior to 20 completed weeks of gestational age.
Stillbirth | after 20 weeks of gestation
  Stillbirth is defined as the death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age including deaths during labor.
Ectopic pregnancy | After 4 to 6 weeks of embryo transfer
  Ectopic pregnancy is defined as a pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Multiple pregnancy | 7 weeks of gestation
  Multiple pregnancy is defined as a pregnancy with two or more gestational sacs or positive heart beats at 7 weeks of gestation.
Gestational diabetes mellitus | At 28 weeks of pregnancy
  Newly diagnosed diabetes or gestational diabetes at 28 weeks of pregnancy confirmed by 75 g oral glucose tolerance test.
hypertensive disorders of pregnancy | From 20 weeks of gestation up to at birth
preterm birth | At birth
  Delivery of a fetus at less than 37 and more than 28 weeks gestational age
low birth weight | At birth
  Weight of baby born < 2500 g
Very low birth weight | At birth
  Weight of baby born < 1500 g
high birth weight | at birth
  Weight of baby born > 4000 g
large for gestational age | at birth
  large for gestational age is defined as birth weight greater than 90th percentile for gestation, based on standardised ethnicity-based charts
small for gestational age | at birth
  small for gestational age is defined as less than 10th percentile for gestational age at delivery based on standardised ethnicity-based charts.
Early neonatal death | within 7days of birth
  Early neonatal death refers to death of a live born baby within 7days of birth
Congenital anomaly | Birth to first year of life
  Any congenital anomalies detected in baby born

CONTACTS AND LOCATIONS:
Overall Officials: Juanzi Shi, Doctor, Study Chair — Center for Reproductive Medicine, Northwest Women's and children's Hospital, Xi'an, shaanxi. china
Locations (1):
- Center for Reproductive Medicine, Northwest Women's and Children's Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No